CLINICAL TRIAL: NCT03382678
Title: CEGIR 7807: Validation of Online Cohort of EGID Patients Enrolled in RDCRN CEGIR Contact Registry
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-5652; 5U54AI117804-03 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Gastrointestinal Disorders
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to validate the online cohort of EGID patients enrolled in the RDCRN CEGIR CR. In order to achieve this objective, the investigators will determine the agreement between self-reported EGID information by the enrollees and their physician's report and medical records. All participants enrolled in the RDCRN CEGIR CR with EGIDs will be invited via email to participate in this study.

DETAILED DESCRIPTION:
All individuals with EGID and enrolled in the RDCRN CEGIR CR will be invited to participate in this survey. As of 04/28, 1567 EGID patients have enrolled in CEGIR CR [EoE=1,217, EG=56, EGE=65, EC=52; multiple diseases=177]

The survey will be conducted through a pre-designed questionnaire. The questionnaire will be sent to participants via an introductory email wherein subjects will be informed about the purpose of this study. The questionnaire will gather self-reported clinical information (such as diagnosis, endoscopic procedures, histological findings in mucosal biopsies, and therapeutic plan). Consent will be obtained from participants to contact their physicians and allow their physicians to share relevant clinical information from their medical records.

Physicians identified by participants will be emailed a website link which will take them to a questionnaire. This questionnaire is designed to gather relevant information as documented in the patient's clinical records. Physicians will be able to submit the information online. It is anticipated that responding to this questionnaire would take less than 10 minutes of their time.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the RDCRN CEGIR Contact Registry, and with Internet access.
* Diagnosis of EGID (EoE, EG, EGE, EE and/or EC)
* Age: all ages. Parents/guardian of children < 18 years of age will respond to the questionnaire on behalf of their child.

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Unaffected family members of EGID patients
* European Union participants who did not complete General Data Protection Regulation requirements.

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with EGID
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Validation of EGID diagnosis | 10 months
  Assess the validity of self-reported EGID diagnosis by comparing to physician reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Rare Diseases Clinical Research Network website — http://www.rarediseasesnetwork.org/cms/CEGIR